CLINICAL TRIAL: NCT05601726
Title: First-In-Human, Open Label, Dose Escalation Study to Evaluate Safety, PK and PD of ABD-3001 As Monotherapy in Relapsed/Refractory Acute Myeloid Leukemia or High/Very-high Risk Myelodysplastic Syndromes Patients, Ineligible for Intensive or New Generation Targeted Therapy.
Brief Title: First-in-human Study Aiming to Characterize the Safety, Tolerability, Pharmacokinetic and Preliminary Signs of Activity of ABD-3001 in Refractory or Relapsed AML and High Risk MDS Adult Patients
Acronym: ODYSSEY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advanced BioDesign (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABD3001CLIN1
Record Dates: First submitted 2022-10-17; First posted 2022-11-01 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia, Adult; Myelodysplastic Syndromes
Keywords: Acute Myeloid Leukemia, Adult; Myelodysplastic syndromes; First in Human; ABD-3001
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — dimethylthioampal

STUDY DESIGN:
Intervention Model Description: This First In Human (FIH) study is a prospective, open-label, multicenter, Phase 1 study, with a dose escalation design, followed by an optimized design. It will consist in a Single Ascending Dose (SAD) part and a Multiple Ascending Dose (MAD) part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Administration Dose (SAD) of ABD-3001 (Experimental): Dose escalation of 6 doses level using a 3+3 design.
  Interventions: Drug: ABD-3001
- Multiple Administration Dose (MAD) of ABD-3001 (Experimental): 3 doses regimens in parallel during 3 cycles of 28 days
  Interventions: Drug: ABD-3001

INTERVENTIONS:
Drug: ABD-3001 — Each patient will receive a fixed 4 hours-intravenous infusion dose of ABD-3001 once or twice a week.
  For SAD : The first dose of the first cohort will receive an estimated infusion dose of 18 mg/m² at Day 1. Subsequent cohorts will be given the following doses: 54 mg/m², 135 mg/m², 270 mg/m², 405 mg/m², 540 mg/m².
  Other Names: DIMATE
  Arms: Single Administration Dose (SAD) of ABD-3001
Drug: ABD-3001 — For MAD :
  Based on all data gathered during the SAD including safety, PK and preliminary efficacy data, up to three doses were selected in accordance with the Safety review Committee (SRC). A dosage optimization analysis was performed at the end of the SAD cohort 6 using population pharmacokinetic modelling to set the optimal frequency of infusion per week for each selected dose to achieve sustained exposition throughout the treatment period. Based on this analysis, the Sponsor, in agreement with the SRC, defined 3 doses regimens that will be set up in parallel, with infusion of ABD-3001 once or twice a week during 3 cycles of 28 days.
  Other Names: DIMATE
  Arms: Multiple Administration Dose (MAD) of ABD-3001

SUMMARY:
This First In Human (FIH) study is a prospective, open-label, multicenter, Phase 1 study, with a dose escalation design, followed by an optimized design. It will consist in a Single Ascending Dose (SAD) part and a Multiple Ascending Dose (MAD) part.

DETAILED DESCRIPTION:
This FIH study combines, in patients with primary refractory or relapsed AML patients and in patients with high risk MDS a Single Ascending Dose (SAD) part (Part A) and a Multiple Ascending Dose (MAD) part (Part B).

The objective of the SAD phase is to explore a wide range of dose administered as a single and fixed 4-hours intravenous infusion in order to select a dose and a dosing frequency (determined using pharmacokinetic and pharmacodynamics parameters).

The objective of the MAD is to elucidate the pharmacokinetic (PK) and pharmacodynamics (PD) of multiple doses of ABD-3001. The dose levels and dosing intervals (i.e., time between consecutive doses) will be selected as those that are predicted to be safe from the SAD. Dose levels and dosing frequency will be derived from data obtained during the SAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory Acute Myeloid Leukemia (AML) after failing at least one therapy regimen and a salvage treatment or are not eligible for salvage treatment regimens including targeted therapy
* Patients with relapsed/refractory Myelodysplastic syndrome (MDS) ineligible for salvage treatment who are diagnosed high-risk and very high-risk using Revised International Prognostic Scoring System (IPSS-R) prognostic risk categorization
* Patients not eligible to alloSCT
* Negative blood or serum/urine pregnancy test

Exclusion Criteria:

* Patients with acute myeloid leukemia (AML) with Inv(16) MYH11-CBF-Beta or t(8;21) AML-ETO RUNX1-RUNX1 or (PML/RARA) karyotype abnormalities and eligible to targeted therapies
* Participants with clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia
* Ongoing immunosuppressive treatment
* Hematopoietic stem cell transplantation (HSCT) performed within 3 months prior to study Visit 1
* Active infection requiring intravenous anti-infectious treatment during the screening period
* Life-threatening illnesses other than the studied one, uncontrolled medical conditions or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety or interfere with the patient's ability to comply with the study activities
* Anti-tumor therapy within 14 days of study Visit 1
* Prior participation in an interventional investigational clinical study (drug or medical device) within 21 days of study Visit 1
* Radiotherapy within 28 days prior to study Visit 1
* Current history of seropositivity to human immunodeficiency virus (HIV) or infection with active hepatitis C virus (HCV) or active hepatitis B virus (HBV) or active SARS-CoV-2 (Covid-19) or Syphilis, or Cytomegalovirus (CMV), or Epstein-Barr virus (EBV), or Human T-Lymphotropic Virus (HTLV1)
* History of other malignancy in the last 12 months prior to study Visit 1
* Other active solid tumor
* Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or Left Ventricular Ejection Fraction (LVEF) <50% attested by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within 28 days of C1D1 prior to study Visit 1 (Day 1, start of study therapy)
* Subjects with a history of myocardial infarction within the last 3 months prior to study Visit 1 (Day 1, start of study therapy)
* Subjects with heart-rate corrected QT (QTc) interval ≥450 ms or other factors that increase the risk of QT prolongation or arrhythmic events
* Major surgery within 4 weeks prior to study Visit 1 (Day 1, start of study therapy)
* Any condition deemed by the investigator to be likely to interfere with a subject's ability to participate in the clinical trial MAD specific exclusion criteria: Patients who have been part of SAD and have experienced a DLT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
SAD : Estimation of the Maximum Tolerated Dose (MTD) of ABD-3001 as well as the doses and frequencies to be explored during the MAD | 7 days for SAD part
  The primary endpoint is to assess the recommended dose range to be tested during the MAD by evaluation of incidence of patients who experienced Dose Limiting Toxicities (DLTs). according to CTCAE v5.0.
  The recommendation for doses to be tested during the MAD will be determined using all available data, which will include Dose Limiting Toxicities (DLTs), MTD if it has been reached, and other toxicities, signs of anti-leukemic activity, pharmacokinetic and pharmacodynamic characteristics.
MAD : To evaluate the safety, tolerability and to define a recommended dose range for further trials. | 3 months for MAD part.
  To assess the impact of ABD-3001 on safety and on its tolerability by evaluating:
  1. Incidence of Adverse Events as characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0 Nov. 27, 2017)), timing, seriousness, and relationship to ABD-3001 either observed by the investigator during physical examination, or reported spontaneously by the patient,
  2. Incidence of laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v5.0 Nov. 27, 2017), and timing.

SECONDARY OUTCOMES:
SAD : To evaluate the overall safety and tolerability profile of ABD-3001 | 7 days for SAD part
  To assess the impact of ABD-3001 on safety and on its tolerability by evaluating:
  1. Incidence of Adverse Events as characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0 Nov. 27, 2017)), timing, seriousness, and relationship to ABD-3001 either observed by the investigator during physical examination, or reported spontaneously by the patient,
  2. Incidence of laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v5.0 Nov. 27, 2017), and timing,
SAD: To assess the pharmacokinetic (PK) parameters of ABD-3001 | 7 days for SAD part
  Maximum concentration (Cmax) of DIMATE and metabolites (CEY1410/H11)
SAD: To assess the pharmacokinetic (PK) parameters of ABD-3001 | 7 days for SAD part
  Time to maximum concentration (Tmax)
SAD: To assess the pharmacokinetic (PK) parameters of ABD-3001 | 7 days for SAD part
  Area Under the plasma Concentration versus time curve (AUC)
SAD: To assess the pharmacokinetic (PK) parameters of ABD-3001 | 7 days for SAD part
  Elimination half-life.
MAD : 1. To assess the pharmacokinetic (PK) parameter of multiple administration of ABD-3001. | 3 months for MAD part.
  PK parameter assessment: maximum concentration (Cmax) of DIMATE and metabolites (CEY1410/H11)
MAD : 2. To assess the pharmacokinetic (PK) parameter of multiple administration of ABD-3001. | 3 months for MAD part.
  PK parameter assessment: time to maximum concentration (Tmax)
MAD : 3. To assess the pharmacokinetic (PK) parameter of multiple administration of ABD-3001. | 3 months for MAD part.
  PK parameter assessment: Area Under the plasma Concentration versus time curve (AUC)
MAD : 4. To assess the pharmacokinetic (PK) parameter of multiple administration of ABD-3001. | 3 months for MAD part.
  PK parameter assessment: elimination half-life.
MAD : 1. To assess the pharmacodynamic (PD) parameter of multiple administration of ABD-3001. | 3 months for MAD part.
  PD parameter assessment: ALDH activity measurement in red blood cells
MAD : 2. To assess the pharmacodynamic (PD) parameter of multiple administration of ABD-3001. | 3 months for MAD part.
  PD parameter assessment: JUNK protein phosphorylation in plasma.
MAD : To evaluate the anti-leukemic activity as assessed by overall response rate (ORR: complete response [CR] + complete response with incomplete hematopoiesis [CRi] + morphologic leukemia-free state [MFLS] + partial response [PR]) | 3 months for MAD part.
  To assess the potential preliminary evidence of anti-leukemia activity at each cycle using response criteria in AML without MRD assessment as defined by ELN 2022
MAD: To evaluate the duration of ORR. | 3 months for MAD part.
  To assess duration of ORR.
MAD: To evaluate Event free survival (EFS) and overall survival (OS) rates at 3-months and 6-months after the end of treatment | 3 months for MAD part.
  To assess the Event Free Survival and the Overall Survival as defined by ELN2022 until 6-months after end of treatment.
MAD: To assess the PRO-QoL during the treatment. | 3 months for MAD part.
  To assess the impact of ABD-3001 on quality of life according QLQ-C30 questionnaire at D1 of each cycle and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BASSET, Study Director — Advanced BioDesign
Locations (3):
- France (3):
  - Hôpital de la Timone, Marseille, France
  - Hôpital Saint-Louis, Paris, France
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venton G, Colle J, Tichadou A, Quessada J, Baier C, Labiad Y, Perez M, De Lassus L, Loosveld M, Arnoux I, Abbou N, Ceylan I, Martin G, Costello R. Reactive oxygen species and aldehyde dehydrogenase 1A as prognosis and theragnostic biomarker in acute myeloid leukaemia patients. J Cell Mol Med. 2024 Oct;28(19):e70011. doi: 10.1111/jcmm.70011. PMID 39392121